CLINICAL TRIAL: NCT06357988
Title: MATCH Treatment Subprotocol T: GDC-0449 (Vismodegib) in Patients With Tumors (Except Basal Cell Skin Carcinoma) With Smoothened (SMO) or Patched 1 (PTCH1) Mutations
Brief Title: Testing GDC-0449 (Vismodegib) as Potentially Targeted Treatment in Cancers With Smoothened or Patched 1 Mutant Tumors (MATCH - Subprotocol T)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01149; NCI-2024-01149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-T (Other: ECOG-ACRIN Cancer Research Group); EAY131-T (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-09; First posted 2024-04-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; Nuclear Medicine Department, Hospital; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Vismodegib) (Experimental): Patients receive vismodegib orally (PO) daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or nuclear study during screening, tumor biopsy on study and CT scan, MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Radionuclide Imaging; Drug: Vismodegib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Radionuclide Imaging — Undergo nuclear study
  Other Names: NM; Nuclear Medicine; nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; Scintigraphy
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449

SUMMARY:
This phase II MATCH treatment trial tests how well GDC-0449 (vismodegib) works for treating patients with solid tumors, lymphoma, or multiple myeloma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that does not respond to treatment (refractory) and who have a smoothened or patched 1 genetic mutation. Vismodegib is a type of medication called a hedgehog signaling pathway antagonist and works by blocks a type of protein involved in tissue growth and repair and may block the growth of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive vismodegib orally (PO) daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or nuclear study during screening, tumor biopsy on study and computed tomography (CT) scan, magnetic resonance imaging (MRI) and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years then every 6 months for year 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must fulfill all eligibility criteria outlined in section 3.1 of MATCH Master protocol (excluding section 3.1.6) at the time of registration to treatment step (step 1, 3, 5, 7)
* Patients must have activating mutations of smoothened (SMO) or deleterious Patched 1 (PTCH1) as determined via the MATCH Master protocol and described in appendix II. See appendix II for information on the smoothened (SMO) or patched 1 (PTCH1) mutations and corresponding levels of evidence
* Patient must not have basal cell carcinoma
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have NONE of the following cardiac criteria:

  * No clinically unstable abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block
  * No factors that increase the risk of corrected QT (QTc) prolongation or risk of arrhythmic events such as congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age
* Patients with known left ventricular dysfunction must have ECHO or nuclear study (multigated acquisition [MUGA] scan or first pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients must not have known hypersensitivity to GDC-0449 (vismodegib) or compounds of similar chemical or biologic composition
* Women of childbearing potential and men who are sexually active must agree to use adequate contraception defined as appropriate double barrier method of birth control (such as female use of a diaphragm, intrauterine device (IUD), sponge and spermicide, in addition to the male use of a condom or involve female use of prescribed "birth control pills" or a prescribed birth control implant). Both double barrier contraception and birth control pills or implants must be used for at least one week prior to the start of the study and continue for 24 months after completion of study for women, and 3 months after completion of study for men

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-02-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 90% two-sided confidence interval is calculated for ORR. For the purposes of this study, patients should be re-evaluated for response:
  * For treatments given in 21 day (3 week) cycles: every 3 cycles (9 weeks) for the first 33 cycles, and every 4 cycles thereafter (12 weeks)
  * For treatments given in 28 day (4 week) cycles: every 2 cycles (8 weeks) for the first 26 cycles, and every three cycles thereafter (12 weeks)
  * For treatments given in 42 day (6 week) cycles: every 2 cycles (12 weeks)

SECONDARY OUTCOMES:
Overall survival (OS) | From start of treatment that step until death, or censored at the date of last contact, assessed up to 3 years
  Will be evaluated specifically for each drug (or step). OS will be estimated using the Kaplan-Meier method.
6-month progression-free survival (PFS) rate | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed at 6 months
  Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Progression free survival | From start of treatment on that step until determination of disease progression or death from any cause, censored at the date of last disease assessment for patients who have not progressed, assessed up to 3 years
  PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm